CLINICAL TRIAL: NCT05073601
Title: Thyroid Gland Dysfunction and Vitamin D Receptor Polymorphism in Keratoconus
Brief Title: Thyroid Gland Dysfunction and Vitamin D Polymorphism in Keratoconus
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Azmy, assistant professor, Mansoura University
Other Study IDs: R.21.01.1157.R1
Record Dates: First submitted 2021-09-22; First posted 2021-10-11 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Keratoconus
Keywords: Thyroid dysfunction; Vitamin D; Polymorphism; keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5ml venous blood was withdrawn from all subjects included in the study; 2ml on ethylenediamine tetraacetic acid (EDTA) for genetic study and 3ml on a plain tube for thyroid hormones and serum 25-(OH) vitamin D measurement. The blood samples for hormonal assessment were centrifuged then serum samples were stored at --20°C till analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: group of subjects with healthy cornea
  Interventions: Diagnostic Test: ELISA,DNA extraction
- keratoconus group: group of keratoconus patients with no history of thyroid dysfunction
  Interventions: Diagnostic Test: ELISA,DNA extraction

INTERVENTIONS:
Diagnostic Test: ELISA,DNA extraction — quantitative measurement of (Thyroid stimulating hormon (TSH), free triiodothyronine (FT3)& Free tetraiodothyronine(FT4)) measured using ELISA . Serum 25-OH vitamin D measured using ELISA. Serum 25-OH vitamin D will be classified based on 2012 American Endocrine Society guidelines into deficient (< 20ng/ml), insufficient ( 21 -30 ng/ml) and sufficient (> 30 ng/ml).vitamin D receptor polymorphisms was done in 3 steps: a) DNA extraction from whole blood using Gene Jet gene DNA Purification kits . b) PCR: three Vitamin D receptor polymorphisms were tested [Taq I (restriction enzymes according to single nucleotide polymorphism ) (rs731236), Apa I (rs7975232) and Bsm I (rs1544410)] using polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP). Genomic DNA was amplified using certain primers

SUMMARY:
This prospective study the thyroid gland dysfunction and vitamin D receptor polymorphism in keratoconus patients

DETAILED DESCRIPTION:
This is a prospective observational study in which blood samples are collected from keratoconus patients looking for thyroid dysfunction and vitamin D levels in the serum and assessing the Vitamin D receptor polymorphism in comparison to healthy control.

ELIGIBILITY:
Inclusion Criteria:

* keratoconus patients without previously diagnosed thyroid disorder in comparison to healthy control without known systemic disease and with normal cornea who were selected from candidates of refractive surgery with normal topography

Exclusion Criteria:

* patients who could not provide informed consent or the necessary samples for any reason, patients with associated other ophthalmic pathologies or systemic disorders were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient clinic of Mansoura ophthalmic center
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
concentration of free T3 | 2month
  pg/ml
concentration of free T4 | 2 month
  ng/dl
concentration of TSH | 2 month
  milli-international units per liter
vitamin D receptor polymorphism | 2 month
  number of participant with vitamin D receptor polymorphism

SECONDARY OUTCOMES:
serum vit D | 2 month
  concentration of Serum 25 OH vitamin D (ng /ml)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Azmy, Principal Investigator — Mansoura University
Locations (1):
- Eman Azmy, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided